CLINICAL TRIAL: NCT05924191
Title: Evaluation of the Preventive Effect of Photobiomodulation in the Postoperative Period of Extractions of Retained Lower Third Molars: a Double-blind Randomized Controlled Study
Brief Title: Preventive Effect of Photobiomodulation in the Postoperative Period of Extractions of Retained Lower Third Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Clinical colaborator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIRUCU
Record Dates: First submitted 2023-06-18; First posted 2023-06-29 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Molar, Third; Photobiomodulation
Keywords: photobiomodulation; corticosteroids; extraction; edema; pain; mouth opening; quality of life; randomized clinical trial
MeSH Terms: conditions — Edema; Pain | interventions — Low-Level Light Therapy; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental group (n=30 surgeries) - the participants will receive the FBM, 1 hour before the surgical procedure, plus a placebo tablet, with the same physical and organoleptic characteristics, composed of corn starch, without harmful effects on health and simulating Dexamethasone (Celsius Laboratory, Montevideo, Uruguay).).
  Interventions: Device: Photobiomodulation; Drug: Placebo Corticosteroid
- Control Group (Active Comparator): Control group (n=30 surgeries) - patients will receive conventional treatment with Dexamethasone 8 mg (Corodex, Laboratorio Celsius, Montevideo, Uruguay) PO 1 hour before surgery (Almeida et al 2019), plus simulation of FBM application. The Laser device will be disconnected and will be applied to the same points as in the experimental group, in the immediate pre-operative period (Baseline).
  Interventions: Device: Simulation Photobiomodulation; Drug: Corticosteroid

INTERVENTIONS:
Device: Photobiomodulation — Intra-oral irradiations wll be performed with a low intensity Laser device at 4 anatomical points, with a wavelength of 660 nm. The extraoral FBM will be applied with 1 cluster (20cm2) with a wavelength of 630nm. Subsequently, the same region will be irradiated with the same cluster, using the 4 LEDs with a wavelength of 850 nm 1 hour before performing the surgery.
  Arms: Experimental Group
Drug: Placebo Corticosteroid — Participants will receive 1 hour before the surgery a placebo tablet, with the same physical and organoleptic characteristics, composed of corn starch, without harmful effects on health and simulating Dexamethasone (Celsius Laboratory, Montevideo, Uruguay).).
  Arms: Experimental Group
Device: Simulation Photobiomodulation — The irradiation simulations will be practiced in the same anatomical points described in the experimental group. This protocol will be carried out 1 hour before the surgical procedure (Baseline). The Laser device will be disconnected and its beep sound will be recorded and run on simulating the irradiation.
  Arms: Control Group
Drug: Corticosteroid — The patients will receive Dexamethasone 8 mg (Corodex, Laboratorio Celsius, Montevideo, Uruguay) PO 1 hour before surgery (Almeida et al 2019)
  Arms: Control Group

SUMMARY:
Third molar extraction is one of the most performed surgical procedures in Dentistry. A comfortable postoperative period and rapid return to daily activities increase the need to control the inflammatory response and its signs and symptoms such as pain, edema, and lockjaw. Therefore, the objective of this study is to evaluate the efficacy of the prophylactic use of Photobiomodulation in the reduction of edema in the postoperative period of extractions of retained lower third molars.The primary study variable will be postoperative edema measured in millimeters, 48 hours after surgery, and the secondary variables will be: pain, lockjaw, local temperature (measured with a thermographic camera), dysphagia, and the need to ingest nonsteroidal analgesics (Acetaminophen)These variables will be evaluated at the beginning of the study (baseline), at 2 and 7 days post-surgery. All adverse effects will be recorded. The data obtained will be represented by their means ± SD and the p value will be set at 0.05.

DETAILED DESCRIPTION:
Third molar extraction is one of the most performed surgical procedures in Dentistry. A comfortable postoperative period and rapid return to daily activities increase the need to control the inflammatory response and its signs and symptoms such as pain, edema, and lockjaw. To control these events, the prophylactic use of anti-inflammatory steroids has been widely recommended by some authors. However, there is no strong evidence on the real benefits of its use as opposed to its possible side effects. Photobiomodulation has proven to be a good alternative when applied in the postoperative period to control pain, edema and lockjaw. On the contrary, its application prior to a procedure of this type has not been sufficiently evaluated. Therefore, the objective of this study is to evaluate the efficacy of the prophylactic use of Photobiomodulation in the reduction of edema in the postoperative period of extractions of retained lower third molars. Healthy individuals (ASA I), who have an indication for extraction and are included in the study, will be randomly divided into two groups: Control Group: with the administration of prophylactic Corticosteroid (Dexamethasone 8 mg/ 1h before surgery), and the simulated application of Photobiomodulation, under the same protocol as the Study Group and Study Group: to which Photobiomodulation will be applied by means of intraoral Low Intensity Laser with wavelengths of 660nm and 808nm applied at 4 anatomical points (power of 0.1W, radiant exposure of 1,061 J/cm2 and energy of 3J per point and an application time of 30 seconds, totaling 12J of energy). Besides, the extraoral application will be carried out with a cluster device of combined LEDs with a total exposure area of 20cm2, which will be composed of 5 LEDs with a wavelength of 630nm (power of 0.25W per LED, a radiant exposure of 3 J /cm2 and energy of 12 J per LED spot, with an exposure time of 48 seconds) and 4 LEDs with a wavelength of 850 nm (power of 0.3W per LED, a radiant exposure of 2.4 J/cm2 and an energy of 12J per LED point, and an exposure time of 40 seconds). The Study Group will be administered a placebo tablet simulating Dexamethasone, also 1 h before the surgical procedure. The primary study variable will be postoperative edema measured in millimeters, 48 hours after surgery, and the secondary variables will be: pain, lockjaw, local temperature (measured with a thermographic camera), dysphagia, and the need to ingest nonsteroidal analgesics (Acetaminophen) after the first 3 postoperative days, where Ketorolac 10 mg will be administered orally, in a regulated manner. These variables will be evaluated at the beginning of the study (baseline), at 2 and 7 days post-surgery. All adverse effects will be recorded. The data obtained will be represented by their means ± SD and the p value will be set at 0.05.

Keywords: photobiomodulation, corticosteroids, extraction, edema, pain, lockjaw, quality of life, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present retained lower third molars, according to the degree of surgical difficulty of the procedure and the anatomical position.The selected molars will be those classified according to classes II and III and/or B or C of Pell and Gregory Classification; in vertical or mesio-angular position, according to the Winter Classification or Class II with need for ostectomy or III, with need for ostectomy and odontosection of the Prant Scale, modified by Amarillas-Escobar et al.
* That have an indication for the extraction of the lower third molars (due to recurrent infections, bad anatomical position, orthodontic indication) or a professional indication presented in writing and that are healthy (ASA I, with a negative medical history).
* Male or female gender.
* Age between 18 and 50 years.
* Good oral hygiene.
* That they agree to participate in the study, after reading and signing the Informed Consent for participation in clinical research.

Exclusion Criteria:

* Carriers of local alterations that contraindicate surgical intervention or complicate the postoperative period (example: acute phase pericoronitis in the last 30 days, ankylosis of the temporomandibular joint).
* Smokers,
* Presenting absence of upper and lower central incisors,
* With a medical history of photosensitivity
* During pregnancy or lactation,
* That they were using anti-inflammatories or analgesics,
* Allergic to any of the drugs used in the research (amoxicillin, ketorolac, acetaminophen, dexamethasone, chlorhexidine 2%, local anesthetics, sodium bisulfite, etc.)
* That during surgery they present any type of complication (bleeding, transoperative difficulties, etc.), because these cases are not included within the expected pattern behavior for this type of surgery (these cases will be reported),
* Surgical time greater than 90 minutes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative Edema baseline | Edema wil be evaluated immediatly before the surgery (baseline)
  To evaluate post-surgical edema (Ustun et al, 2003, Mello et al, 2001), 3 measurements will be determined on the patient's face, with a malleable tape measure graduated in mm (millimeters), previously sanitized, as follows: tragus-pogonion; tragus- labial commissure and mandibular angle (gonion)- external corner of the eye (external canthus). The reference points will be marked with indelible dermographic ink and will remain unchanged throughout the post-surgical evaluation period, for this purpose The patient will be asked to ensure the unaltered conservation of those points
Postoperative Edema - 48 hours postoperative | Edema wil be evaluated at 2 postoperative days.
  To evaluate post-surgical edema (Ustun et al, 2003, Mello et al, 2001), 3 measurements will be determined on the patient's face, with a malleable tape measure graduated in mm (millimeters), previously sanitized, as follows: tragus-pogonion; tragus- labial commissure and mandibular angle (gonion)- external corner of the eye (external canthus). The reference points will be marked with indelible dermographic ink and will remain unchanged throughout the post-surgical evaluation period, for this purpose The patient will be asked to ensure the unaltered conservation of those points.
Postoperative Edema - 7day postoperative | Edema wil be evaluated at 7 postoperative days.
  To evaluate post-surgical edema (Ustun et al, 2003, Mello et al, 2001), 3 measurements will be determined on the patient's face, with a malleable tape measure graduated in mm (millimeters), previously sanitized, as follows: tragus-pogonion; tragus- labial commissure and mandibular angle (gonion)- external corner of the eye (external canthus). The reference points will be marked with indelible dermographic ink and will remain unchanged throughout the post-surgical evaluation period, for this purpose The patient will be asked to ensure the unaltered conservation of those points.

SECONDARY OUTCOMES:
Postoperative Pain baseline | In this study, the VAS will be used immediately before surgery (Baseline)
  Pain sensitivity - The Visual Analogue Scale (VAS) is the most commonly used instrument for the assessment of postoperative pain in oral surgeries when FBM is used as post-surgical palliative therapy (Yüksek, Eroglu 2021, Momeni et al 2021, Amarillas -Escobar et al 2010, López-Ramírez et al 2011, Brignardello-Petersen et al 2012, Sierra et al 2013, Sierra et al 2015).
  A rule will be used, graduated in cm, 10 cm long. One of the extremes represents "0", which means "no pain" and the other represents "10" which indicates "unbearable pain". The intermediate graduation gives patients the possibility of rating the intensity of their painful experience, from 0 to 10. This rule will be the same for all study participants and the indications for its use and marking will be given to the patient, always by the same operator
Postoperative Pain - 48 hours | In this study, the VAS will be used at 2 postoperative days
  Pain sensitivity - The Visual Analogue Scale (VAS) is the most commonly used instrument for the assessment of postoperative pain in oral surgeries when FBM is used as post-surgical palliative therapy (Yüksek, Eroglu 2021, Momeni et al 2021, Amarillas -Escobar et al 2010, López-Ramírez et al 2011, Brignardello-Petersen et al 2012, Sierra et al 2013, Sierra et al 2015).
  A rule will be used, graduated in cm, 10 cm long. One of the extremes represents "0", which means "no pain" and the other represents "10" which indicates "unbearable pain". The intermediate graduation gives patients the possibility of rating the intensity of their painful experience, from 0 to 10. This rule will be the same for all study participants and the indications for its use and marking will be given to the patient, always by the same operator
Postoperative Pain - 7 days | In this study, the VAS will be used 7 days before surgery
  Pain sensitivity - The Visual Analogue Scale (VAS) is the most commonly used instrument for the assessment of postoperative pain in oral surgeries when FBM is used as post-surgical palliative therapy (Yüksek, Eroglu 2021, Momeni et al 2021, Amarillas -Escobar et al 2010, López-Ramírez et al 2011, Brignardello-Petersen et al 2012, Sierra et al 2013, Sierra et al 2015).
  A rule will be used, graduated in cm, 10 cm long. One of the extremes represents "0", which means "no pain" and the other represents "10" which indicates "unbearable pain". The intermediate graduation gives patients the possibility of rating the intensity of their painful experience, from 0 to 10. This rule will be the same for all study participants and the indications for its use and marking will be given to the patient, always by the same operator
Postoperative use of analgesics - baseline | The amount of analgesics will be recorded in the baseline.
  Amount of analgesics necessarily ingested, as a rescue: The amount of analgesic (Acetaminophen), a drug with a purely analgesic effect (Józwiak-Bebenista 2014) ingested by the patient (500 mg every 6 hours if the pain continues), will be recorded. At the beginning of the investigation, each patient will be given a form to record daily consumption, after the 3rd. post-operative day, and must be kept until the end of its use, at surgical discharge. At the end of the study, the amount of Acetaminophen tablets used will be evaluated as a secondary variable. The adherence of the participants to the study will be monitored through this means, asking the patients to present the form to verify its use.
Postoperative use of analgesics - 7th days | The amount of analgesics will be recorded after the third postoperative day until the 7th. post-operative day.
  Amount of analgesics necessarily ingested, as a rescue: The amount of analgesic (Acetaminophen), a drug with a purely analgesic effect (Józwiak-Bebenista 2014) ingested by the patient (500 mg every 6 hours if the pain continues), will be recorded. At the beginning of the investigation, each patient will be given a form to record daily consumption, after the 3rd. post-operative day, and must be kept until the end of its use, at surgical discharge. At the end of the study, the amount of Acetaminophen tablets used will be evaluated as a secondary variable. The adherence of the participants to the study will be monitored through this means, asking the patients to present the form to verify its use.
Postoperative Trismus - baseline | In the present study, the previously calibrated evaluators will measure the mouth opening in each patient before the surgeries (baseline)
  Evaluation of post-operative trismus- Spasms in the masticatory muscles (lockjaw) can limit or even prevent the normal opening of the mouth after surgical removal of impacted lower third molars (Yüksek, Eroğlu, 2021, López-Ramírez et al ., 2012; Aras; Güngörmüs, 2009; Aras; Güngörmüs, 2010; Amarillas-Escobar et al., 2010; Ferrante et al., 2013). This result is generally evaluated by measuring the distance between the incisal edges of the upper and lower central incisors, using a caliper, graduated in mm (millimeters) (Yüksek, Eroğlu, 2021, Sampaio-Filho et al., 2017 , Bauer et al. 2013).
Postoperative Trismus 48 hours | In the present study, the previously calibrated evaluators will measure the mouth opening in each patient at 2 postoperative days.
  Evaluation of post-operative trismus- Spasms in the masticatory muscles (lockjaw) can limit or even prevent the normal opening of the mouth after surgical removal of impacted lower third molars (Yüksek, Eroğlu, 2021, López-Ramírez et al ., 2012; Aras; Güngörmüs, 2009; Aras; Güngörmüs, 2010; Amarillas-Escobar et al., 2010; Ferrante et al., 2013). This result is generally evaluated by measuring the distance between the incisal edges of the upper and lower central incisors, using a caliper, graduated in mm (millimeters) (Yüksek, Eroğlu, 2021, Sampaio-Filho et al., 2017 , Bauer et al. 2013).
Postoperative Trismus - 7 days | In the present study, the previously calibrated evaluators will measure the mouth opening in each patient after 7 postoperative days.
  Evaluation of post-operative trismus- Spasms in the masticatory muscles (lockjaw) can limit or even prevent the normal opening of the mouth after surgical removal of impacted lower third molars (Yüksek, Eroğlu, 2021, López-Ramírez et al ., 2012; Aras; Güngörmüs, 2009; Aras; Güngörmüs, 2010; Amarillas-Escobar et al., 2010; Ferrante et al., 2013). This result is generally evaluated by measuring the distance between the incisal edges of the upper and lower central incisors, using a caliper, graduated in mm (millimeters) (Yüksek, Eroğlu, 2021, Sampaio-Filho et al., 2017 , Bauer et al. 2013).
Postoperative Local temperature baseline | baseline
  Local temperature -To evaluate it a thermographic photograph of the facial skin in the operated area will be taken using a FLIR C5sc 9 camera (Teledyne FLIR, Wilsonville, Oregon, USA). . The quantification of the temperature will be carried out by means of the FLIR Research IR thermal analysis software. In all photographic records, the camera-patient distance will be kept constant, as will the ambient temperature of the place where the thermographic records are made.
Postoperative Local temperature 48 hours | Thermographic photographs wil be taken 2 days after surgery.
  Local temperature -To evaluate it a thermographic photograph of the facial skin in the operated area will be taken using a FLIR C5sc 9 camera (Teledyne FLIR, Wilsonville, Oregon, USA). . The quantification of the temperature will be carried out by means of the FLIR Research IR thermal analysis software. In all photographic records, the camera-patient distance will be kept constant, as will the ambient temperature of the place where the thermographic records are made.
Postoperative Local temperature - 7 days | Thermographic photographs wil be taken 7 days after surgery.
  Local temperature -To evaluate it a thermographic photograph of the facial skin in the operated area will be taken using a FLIR C5sc 9 camera (Teledyne FLIR, Wilsonville, Oregon, USA). . The quantification of the temperature will be carried out by means of the FLIR Research IR thermal analysis software. In all photographic records, the camera-patient distance will be kept constant, as will the ambient temperature of the place where the thermographic records are made.
Postoperative Quality of life - baseline | Quality of life will be evaluated in the baseline
  Impact of the surgical procedure on the quality of life of patients - Two previously calibrated evaluators will ask patients to answer YES or NO to the following 10 questions, as described by Colorado- Bonin et al., 2006; Sato et al., 2009; savin; Grossi et al., 2007, Sierra et al. 2013, Sierra et al. 2015.
  1. Are you maintaining your social activities normally?
  2. Are you working and/or studying normally?
  3. Are you maintaining a normal diet?
  4. Do you have difficulty swallowing because of the surgery?
  5. Do you have difficulty perceiving the taste of food?
  6. Can you chew on the operated side?
  7. Do you have difficulty sleeping because of the surgery?
  8. Do you have difficulty speaking because of the surgery?
  9. Has your physical appearance changed because of the surgery?
  10. Are you angry about the surgery?
Postoperative Quality of life - 48 hours | Quality of life will be evaluated two days after surgery,
  Impact of the surgical procedure on the quality of life of patients - Two previously calibrated evaluators will ask patients to answer YES or NO to the following 10 questions, as described by Colorado- Bonin et al., 2006; Sato et al., 2009; savin; Grossi et al., 2007, Sierra et al. 2013, Sierra et al. 2015.
  1. Are you maintaining your social activities normally?
  2. Are you working and/or studying normally?
  3. Are you maintaining a normal diet?
  4. Do you have difficulty swallowing because of the surgery?
  5. Do you have difficulty perceiving the taste of food?
  6. Can you chew on the operated side?
  7. Do you have difficulty sleeping because of the surgery?
  8. Do you have difficulty speaking because of the surgery?
  9. Has your physical appearance changed because of the surgery?
  10. Are you angry about the surgery?
Postoperative Quality of life - 7 days | Quality of life will be evaluated seven days after surgery,
  Impact of the surgical procedure on the quality of life of patients - Two previously calibrated evaluators will ask patients to answer YES or NO to the following 10 questions, as described by Colorado- Bonin et al., 2006; Sato et al., 2009; savin; Grossi et al., 2007, Sierra et al. 2013, Sierra et al. 2015.
  1. Are you maintaining your social activities normally?
  2. Are you working and/or studying normally?
  3. Are you maintaining a normal diet?
  4. Do you have difficulty swallowing because of the surgery?
  5. Do you have difficulty perceiving the taste of food?
  6. Can you chew on the operated side?
  7. Do you have difficulty sleeping because of the surgery?
  8. Do you have difficulty speaking because of the surgery?
  9. Has your physical appearance changed because of the surgery?
  10. Are you angry about the surgery?
Postoperative Dysphagia baseline | Dysphagia will be evaluated at baseline
  Dysphagia - The evaluation of dysphagia will be carried out through a questionnaire (Sampaio-Filho et al., 2017) that will classify on a numerical scale as follows:
  (0)= total absence of dysphagia.
  1. = dysphagia to solid foods.
  2. = dysphagia to any food, liquid or solid.
Postoperative Dysphagia 48 hours | Dysphagia will be evaluated at 2 days post-surgery
  Dysphagia - The evaluation of dysphagia will be carried out through a questionnaire (Sampaio-Filho et al., 2017) that will classify on a numerical scale as follows:
  (0)= total absence of dysphagia.
  1. = dysphagia to solid foods.
  2. = dysphagia to any food, liquid or solid.
Postoperative Dysphagia - 7 days | Dysphagia will be evaluated 7 days post-surgery
  Dysphagia - The evaluation of dysphagia will be carried out through a questionnaire (Sampaio-Filho et al., 2017) that will classify on a numerical scale as follows:
  (0)= total absence of dysphagia.
  1. = dysphagia to solid foods.
  2. = dysphagia to any food, liquid or solid.
Postoperative Hematoma/ecchymosis - baseline | Hematoma/ecchymosis will be evaluated at baseline
  The presence of hematoma/ecchymosis will be evaluated by measuring the largest diameter of the colorimetric changes in the skin of the jugal and submandibular region with a millimetric graduated malleable rule. The measurement will be carried out by the previously calibrated evaluator, who will classify the appearance of this finding into 4 categories:
  1. non-existent;
  2. the largest diameter is less than 4 cm;
  3. the largest diameter is between 4 and 10 cm;
  4. the largest diameter is greater than 10 cm; as described by Bjornsson et al., (2003).
Postoperative Hematoma/ecchymosis | Hematoma/ecchymosis will be evaluated 2 days after surgery,
  The presence of hematoma/ecchymosis will be evaluated by measuring the largest diameter of the colorimetric changes in the skin of the jugal and submandibular region with a millimetric graduated malleable rule. The measurement will be carried out by the previously calibrated evaluator, who will classify the appearance of this finding into 4 categories:
  1. non-existent;
  2. the largest diameter is less than 4 cm;
  3. the largest diameter is between 4 and 10 cm;
  4. the largest diameter is greater than 10 cm; as described by Bjornsson et al., (2003).
Postoperative Hematoma/ecchymosis - 7 days | Hematoma/ecchymosis will be evaluated 7 days after surgery,
  The presence of hematoma/ecchymosis will be evaluated by measuring the largest diameter of the colorimetric changes in the skin of the jugal and submandibular region with a millimetric graduated malleable rule. The measurement will be carried out by the previously calibrated evaluator, who will classify the appearance of this finding into 4 categories:
  1. non-existent;
  2. the largest diameter is less than 4 cm;
  3. the largest diameter is between 4 and 10 cm;
  4. the largest diameter is greater than 10 cm; as described by Bjornsson et al., (2003).

CONTACTS AND LOCATIONS:
Locations (1):
- Kristianne Porta Santos Fernandes, São Paulo, São Paulo, Brazil